CLINICAL TRIAL: NCT02560805
Title: Post-Traumatic Stress Disorder and Cardiovascular Disease Risk: Role of Sympathetic Overactivity and Angiotensin II
Brief Title: Role of Sympathetic Overactivity and Angiotensin II in PTSD and CV
Acronym: ANG-P
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment and study activities are temporarily suspended due to COVID-19.
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jeanie Park, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00082400
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Nitroprusside; Phenylephrine; Losartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

ARMS (6):
- Veterans with Post-traumatic Stress Disorder (PTSD) (Experimental): For examining Objective 1 of this study, participants with post-traumatic stress disorder (PTSD) will be evaluated using microneurography, static handgrip exercise, cold pressor test, combat virtual reality video clip, and baroreflex sensitivity using sodium nitroprusside and phenylephrine. For the second phase, they will be randomized to either losartan or atenolol.
  Interventions: Procedure: Microneurography; Behavioral: Combat virtual reality video clip; Procedure: Handgrip Exercise; Procedure: Cold Pressor Test (CPT); Drug: Sodium Nitroprusside (SNP); Drug: Phenylephrine
- Control (Experimental): For examining Objective 1 of this study, healthy controls will be evaluated using microneurography, static handgrip exercise, cold pressor test, combat virtual reality video clip, and baroreflex sensitivity using sodium nitroprusside and phenylephrine.
  Interventions: Procedure: Microneurography; Behavioral: Combat virtual reality video clip; Procedure: Handgrip Exercise; Procedure: Cold Pressor Test (CPT); Drug: Sodium Nitroprusside (SNP); Drug: Phenylephrine
- Losartan (Experimental): Participants with PTSD randomized to receive losartan for 8 to 14 weeks.
  Interventions: Drug: Losartan
- Atenolol (Active Comparator): Participants with PTSD randomized to receive atenolol for 8 to 14 weeks.
  Interventions: Drug: Atenolol
- Transcutaneous Vagal Nerve Stimulation (tVNS) (Experimental): Participants with PTSD randomized to receive treatment with tVNS for 8 to 14 weeks.
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)
- Sham Transcutaneous Vagal Nerve Stimulation (tVNS) (Sham Comparator): Participants with PTSD randomized to receive treatment with sham-tVNS for 8 to 14 weeks.
  Interventions: Device: Sham Transcutaneous Vagal Nerve Stimulation (tVNS)

INTERVENTIONS:
Procedure: Microneurography — Skin will be stimulated with a pencil-shaped electrode to find a certain nerve. Once the nerve is found, two tiny sterile wire needles (about the size of acupuncture needles) will be put in the skin. One needle is put just under the skin at a short distance away from the nerve, and the other one into the nerve. The needles are attached to a computer recorder to record the nerve activity. It may take up to one hour to get the needles in the right place. After the tiny needle is in the right place, investigators record nerve activity at rest for about 10 minutes. Then, it will be recorded throughout the rest of the visit (up to 4 hours).
  Arms: Control; Veterans with Post-traumatic Stress Disorder (PTSD)
Behavioral: Combat virtual reality video clip — Subjects will watch a video clip of combat on a computer screen or wearing video goggles.
  Arms: Control; Veterans with Post-traumatic Stress Disorder (PTSD)
Procedure: Handgrip Exercise — Subjects will squeeze a hand dynamometer intermittently.
  Arms: Control; Veterans with Post-traumatic Stress Disorder (PTSD)
Procedure: Cold Pressor Test (CPT) — Subjects' hand will be submerged in cold water (~0-1°C) up to the wrist for 1 minute.
  Arms: Control; Veterans with Post-traumatic Stress Disorder (PTSD)
Drug: Sodium Nitroprusside (SNP) — Subjects will receive sodium nitroprusside 100 µg, which is bolused through an antecubital intravenous catheter.
  Other Names: Nitropress
  Arms: Control; Veterans with Post-traumatic Stress Disorder (PTSD)
Drug: Phenylephrine — Subjects will receive phenylephrine 150 µg, which is bolused through an antecubital intravenous catheter 60 seconds after the sodium nitroprusside bolus
  Arms: Control; Veterans with Post-traumatic Stress Disorder (PTSD)
Drug: Losartan — Losartan will be administered as 25 mg taken orally, once a day for to 8 to 14 weeks.
  Other Names: Cozaar
  Arms: Losartan
Drug: Atenolol — Atenolol will be administered as 25 mg taken orally, once a day for to 8 to 14 weeks.
  Other Names: Tenormin
  Arms: Atenolol
Device: Transcutaneous Vagal Nerve Stimulation (tVNS) — Transcutaneous vagal nerve stimulation (tVNS) is administered using the gammaCore (ElectroCore) TENS device. The gammaCore device is a multi-use, hand-held, rechargeable portable device consisting of a rechargeable battery, signal generating and amplifying electronics, and two buttons to power on the device and for operator control of the stimulation intensity (range 0-40). A small amount of conductive gel is applied to the pair of stainless steel round discs on the device are placed vertically on the skin with the gel. The stimulation is increased until there is a strong vibration and slight muscle contraction in the lower face or neck (usual intensity 15-25). Then the dose is delivered for 2 minutes on the left side of the neck, and on the right side of the neck, for a total of 4 minutes of treatment. Participants will be instructed on the usage of the device and will self-administer up to 4 treatments twice per day.
  Other Names: ElectroCore
  Arms: Transcutaneous Vagal Nerve Stimulation (tVNS)
Device: Sham Transcutaneous Vagal Nerve Stimulation (tVNS) — A sham device that is identical to the gammaCore device will be provided to participants. Participants will be instructed on the usage of the device and will self-administer up to 4 treatments twice per day.
  Arms: Sham Transcutaneous Vagal Nerve Stimulation (tVNS)

SUMMARY:
The purpose of this study is to find out why patients with post-traumatic stress disorder (PTSD) have an increased risk for heart disease and high blood pressure later in life. A second purpose is to find out what causes PTSD patients to have high adrenaline levels during stress. This study will also test if a medicine called losartan improves high adrenaline levels in patients with PTSD and if a certain gene that has to do with high blood pressure might be associated with high adrenaline levels.

DETAILED DESCRIPTION:
More than 2,000,000 soldiers have been deployed to Iraq and Afghanistan in the past decade as part of Operation Enduring Freedom/ Operation Iraqi Freedom/ Operation New Dawn (OEF/OIF/OND), and are returning with high rates of post-traumatic stress disorder (PTSD). The prevalence of PTSD in OEF/OIF/OND veterans is estimated at around 11.5-19.9% post deployment, with prevalence rates of 12.1% and 30.9% in older veterans from the Gulf War and Vietnam era, respectively. PTSD is also common in the general population, as 7% of the US population will meet the diagnostic criteria for PTSD in their lifetime. With these extensive and ongoing conflicts, and the tremendous deleterious mental health and socioeconomic impact of PTSD, research to understand and treat all aspects of PTSD is vitally important.

One less recognized but highly significant consequence of PTSD is an increased risk of hypertension, cardiovascular (CV) disease, and its risk factors. One mechanism likely underlying increased CV risk in PTSD is chronic overactivation of the sympathetic nervous system (SNS). SNS overactivity leads to increased CV risk by increasing blood pressure (BP), and also via BP-independent effects including vascular inflammation, insulin resistance, and myocardial fibrosis.

Chronic inflammation is likely a key culprit contributing to SNS overactivation and blunted baroreflex sensitivity (BRS) in PTSD. In Objective 1 of this study, the researchers will ascertain that humans with PTSD have chronic overactivation of muscle sympathetic nerve activity (MSNA), blunted BRS, and elevated inflammation both at rest and during mental stress.

In addition to chronic inflammation, trauma-related stress is known to activate the renin-angiotensin system (RAS) leading to higher brain angiotensin II (ATII) that is an important mediator of brain inflammation and has a direct sympathoexcitatory effect. Previous studies in both animals and humans with a variety of chronic diseases such as obesity, heart failure, and chronic kidney disease, have shown that blockade of the ATII receptor using angiotensin receptor blockers (ARBs) reduces SNS activity and improves BRS. The extent to which ARB treatment influences SNS activation, BRS, and inflammation in PTSD patients remains unknown. Currently, peripheral sympatholytics such as β-blockers and α-blockers are often prescribed for PTSD symptoms; however, treatment is often complicated by adverse effects including hypotension, orthostasis, fatigue, and erectile dysfunction. In addition, these peripheral sympatholytics cause a reflex increase in central sympathetic output as evidenced by increased MSNA; therefore, these medications may actually contribute to increased CV risk in PTSD. As opposed to peripheral sympatholytics, losartan is well tolerated, without metabolic side effects, and reduces central SNS activation which has potential to impact future CV risk.

Vagal nerve stimulation has been shown in both animal and human studies to safely and effectively reduce sympathetic activity and inflammation. tVNS is a noninvasive method that involves placing a device over the skin overlying the vagus nerve on the neck. The device delivers mild electrical stimulation, using transcutaneous electrical nerve stimulation (TENS) unit. Prior studies have shown that transcutaneous vagal nerve stimulation safely and effectively reduced muscle sympathetic nerve activity in healthy humans and improved heart rate variability, indicating a decrease in sympathetic nervous system (SNS) activity, and a shift in cardiac autonomic function toward parasympathetic (PNS) predominance. Another study, found that tVNS acutely improved cardiac baroreflex sensitivity. Since PTSD patients have high SNS, low PNS activity and impaired baroreflex sensitivity, tVNS may be one safe and noninvasive method of improving autonomic function in this patient population. The researchers will test whether tVNS leads to both an acute and sustained improvement in SNS function in PTSD.

Study Objective 2 evaluates the clinical utility of losartan treatment on autonomic control in humans with PTSD. Participants with PTSD will be randomized to treatment with the ARB losartan (25 mg daily) versus the comparison drug atenolol (25 mg daily) for 8-14 weeks. Alternatively, participants with PTSD may be randomized to treatment with tVNS versus sham-tVNS for 8-14 weeks

ELIGIBILITY:
Inclusion Criteria:

* veterans ages 18-65 years old with PTSD and without PTSD (controls) matched for age, gender, and race.

Exclusion Criteria:

* pregnancy
* hypertension
* diabetes
* heart or vascular disease
* illicit drug use
* excessive alcohol use (>2 drinks per day)
* hyperlipidemia
* autonomic dysfunction
* current treatment with clonidine, beta blockers, angiotensin-converting-enzyme (ACE) inhibitors, or angiotensin II receptor blockers (ARBs)
* treatment with monoamine oxidase (MAO) inhibitors within the last 14 days
* any serious systemic disease
* chronic kidney disease defined as estimated glomerular filtration rate (GFR) < 60 cc/min
* hyperkalemia (serum potassium > 5 meq/dL)
* systolic blood pressure < 100 mm Hg
* diastolic blood pressure < 60 mm Hg
* heart rate < 50 beats/min
* known hypersensitivity to ARBs or beta blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Sympathetic Nerve Activity (MSNA) | Baseline, after study intervention (up to 14 weeks)
  Multiunit postganglionic sympathetic nerve activity is recorded from a tungsten microelectrode inserted into the peroneal nerve with a reference microelectrode inserted in close proximity. Efferent nerve signals are amplified, filtered, rectified and integrated (time constant 0.1 s) to obtain a mean voltage display of MSNA. MSNA bursts are automatically detected using the following criteria: burst-to-noise ratio of 3:1 within a 0.5-s search window, with an average latency of 1.2-1.3 s in burst occurrence from the previous R-wave. MSNA is expressed as burst frequency measured a bursts per minute. MSNA will be examined at rest and during mental stress.

SECONDARY OUTCOMES:
Change in Baroreflex Sensitivity (BRS) | Baseline, after study intervention (up to 14 weeks)
  Afferent sympathetic baroreflex input travels to the brainstem via the glossopharyngeal and vagus nerves and integrate with brainstem centers that regulate efferent SNS (sympathetic BRS) and parasympathetic (cardiovagal BRS) outflow. BRS is defined as the change in interbeat interval (IBI) in milliseconds per unit change in BP. For example, when the BP rises by 10 mmHg and IBI increases by 100 ms, BRS would be 100/10 = 10 ms/mmHg. BRS will be examined at rest and during mental stress.
C-reactive protein (CRP) | Baseline, after study intervention (up to 14 weeks)
  The inflammatory biomarker CRP increases when inflammation is present.
Interleukin 2 (IL-2) | Baseline, after study intervention (up to 14 weeks)
  The inflammatory biomarker IL-2 will be assessed.
Interleukin 6 (IL-6) | Baseline, after study intervention (up to 14 weeks)
  Plasma concentration of the inflammatory biomarker IL-6 will be assessed. IL-6 is increased during injury or illness.
Angiotensin II (ATII) | Baseline, after study intervention (up to 14 weeks)
  ATII will be assessed to determine if ATII signaling contributes to SNS overactivity in PTSD.
Lipoprotein-associated Phospholipase A2 Mass (Lp-PLA2) | Baseline, after study intervention (up to 14 weeks)
  Lp-PLA2 is a unique inflammatory biomarker that is involved in early atherogenesis, endothelial dysfunction, and vascular wall inflammation, which may be elevated in PTSD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No